CLINICAL TRIAL: NCT04969315
Title: Phase I/II First-in-Human Study of TT-10 (PORT-6), an Adenosine 2A Receptor Antagonist, and PORT-7, an Adenosine 2B Receptor Antagonist, as Single Agents and in Combination in Participants With Advanced Selected Solid Tumors
Brief Title: TT-10 (PORT-6) and TT-4 (PORT-7) as Single Agents and in Combination in Subjects With Advanced Selected Solid Tumors
Acronym: ADPORT-601
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Portage Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT-10-101/ADPORT-601; TT-10-101 (Other: Tarus Therapeutics, Inc.); TT-4-101 (Other: Tarus Therapeutics, Inc.)
Record Dates: First submitted 2021-07-05; First posted 2021-07-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Cancer; Castrate Resistant Prostate Cancer; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Cancer (CRC); Endometrial Cancer; Ovarian Cancer
Keywords: Failed or not eligible for standard of care; Advanced Selected Solid Tumors; TT-10; Adenosine; Adenosine Antagonist; A2A; A2AR Inhibitor; PORT-6; ADPORT-601; TT-4; PORT-7; A2B; Dual; A2AR; A2BR
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Dose Escalation (Experimental): Drug: TT-10 (A2A Receptor Antagonist)
  * Supplied in capsules for daily oral administration twice a day (BID)
  * One cycle is considered 28 days
  * Ascending Dose levels are being explored
    * Dose Level 1
    * Dose Level 2
    * Dose Level 3
    * Dose Level 4* *Additional dose levels may be explored, if appropriate based on emerging safety, PK or pharmacodynamic data
  Interventions: Drug: TT-10
- Cohort B: Dose Escalation (Experimental): Drug: TT-4 (A2B Receptor Antagonist)
  * Supplied in capsules for daily oral administration once a day (QD)
  * One cycle is considered 28 days
  * Ascending Dose levels are being explored
    * Dose Level 1
    * Dose Level 2
    * Dose Level 3*
    * *Additional dose levels or frequency may be explored, if appropriate based on emerging safety, PK or pharmacodynamic data
  Interventions: Drug: TT-4
- Cohort C: Dose Escalation (Experimental): Drugs: TT-10 + TT-4 - Dual Receptor Antagonists
  * Both drugs will be supplied in capsules for daily oral administration and administered separately.
  * One cycle is considered 28 days
  * Ascending Dose levels of both drugs are being explored and will be determined after safety review of Cohorts A and B
  Interventions: Drug: TT-10; Drug: TT-4

INTERVENTIONS:
Drug: TT-10 — TT-10 orally administered BID
  Arms: Cohort A: Dose Escalation; Cohort C: Dose Escalation
Drug: TT-4 — TT-4 is orally administered QD
  Arms: Cohort B: Dose Escalation; Cohort C: Dose Escalation

SUMMARY:
The goal of this clinical trial is to evaluate TT-10, TT-4 and TT-10 + TT-4, (Dual Blockade) in participants with advanced selected solid tumors, who have failed or are not eligible for standard of care. The main questions it aims to answer are:

1. To evaluate the safety and tolerability of TT-10, TT-4 and TT-10 + TT-4, (Dual Blockade)
2. To determine the maximum tolerated dose or the recommended phase 2 dose of TT-10, TT-4 and TT-10 + TT-4, (Dual Blockade)
3. To obtain a preliminary estimate of efficacy of TT-10, TT-4 and TT-10 + TT-4, (Dual Blockade) in advanced solid tumors.

DETAILED DESCRIPTION:
Multicenter, open-label dose-escalation Phase I/II clinical study, designed to evaluate the safety, tolerability, PK, PD, anti-tumor activity, and efficacy of TT-10, TT-4 and TT-10 + TT-4 (Dual Blockade).

The Phase Ia portion of the study study will consist of three dose escalation cohorts, to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D), safety and tolerability of TT-10, TT-4, TT-10 + TT-4 and will be conducted in participants with the following advanced cancers:

Cohort A (TT-10): Renal cell cancer (RCC), castrate resistant prostate cancer (CRPC), non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN); who have failed or are not eligible for standard of care treatment.

Cohort B (TT-4): Castrate resistant prostate cancer (CRPC), non-small cell lung cancer (NSCLC), colorectal cancer (CRC), endometrial cancer (EC) and ovarian cancer (OC); who have failed or are not eligible for standard of care treatment.

Cohort C (TT-10 + TT-4): Tumor types from both cohorts will be included and prioritized based on the data observed.

ELIGIBILITY:
To be eligible for inclusion in the dose escalation cohorts or expansion cohorts in this study, participants must meet all of the following criteria:

1. Participants must be ≥18 years of age.
2. Participants or their legal representative must be able to provide written informed consent to participate in the study prior to the performance of any study-specific procedures.
3. Diagnosis of histologically or cytologically confirmed advanced selected solid tumors:

   Cohort A - TT-10 dose escalation:
   1. RCC: Participants with locally advanced or metastatic RCC that have previously received at least two prior systemic regimens, including vascular endothelial growth factor (VEGF)-targeted therapy and checkpoint inhibitor therapy
   2. CRPC: Participants with metastatic CRPC who have previously received a second-generation hormonal agent (unless contraindicated) and a taxane-based chemotherapy.
   3. SCCHN: Participants with advanced or metastatic SCCHN that is incurable by surgery or radiotherapy and that has progressed during or after a platinum-based chemotherapy and/or checkpoint inhibitor therapy (separately or in combination)
   4. NSCLC: Participants with metastatic NSCLC that is intolerant or resistant to standard therapy or for which no standard therapy is available

   Cohort B - TT-4 dose escalation:
   1. CRC: Participants with metastatic CRC that is intolerant or resistant to standard therapy or for which no standard therapy is available
   2. CRPC: Participants with metastatic CRPC who have previously received a second-generation hormonal agent (unless contraindicated) and a taxane-based chemotherapy
   3. NSCLC: Participants with metastatic NSCLC that is intolerant or resistant to standard therapy or for which no standard therapy is available
   4. Endometrial cancer: Participants with metastatic endometrial cancer that is intolerant or resistant to standard therapy or for which no standard therapy is available
   5. Ovarian cancer: Participants with metastatic ovarian cancer that is intolerant or resistant to standard therapy or for which no standard therapy is available

   Cohort C- TT-10 + TT- 4 dose escalation and expansion:

   a. The tumor types will include 1 or more of those enrolled in the respective Escalation Cohorts (A and B), and will be determined following review of the dose escalation data by the SMC.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0 - 1
5. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   a. Participants with CRPC who have metastatic disease that is non-measurable are eligible if screening PSA ≥ 2.0 ng/mL and with Sponsor approval
6. Failure to respond to standard therapy, or for whom no appropriate therapies are available (based on the judgment of the investigator)
7. Consent to baseline biopsy, with the following exceptions:

   1. Participants whose only site(s) of disease are in areas considered moderate or high risk may be enrolled without a fresh biopsy with Sponsor approval;
   2. Archival tissue may be submitted in lieu of a fresh biopsy if collected within 6 months of screening and without intervening systemic therapy.
8. Participants must have adequate hematologic function based on the following:

   * ANC ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
9. Participants must have adequate hepatic function based on the following:

   * Total bilirubin < 1.5 x upper limit of normal (ULN) (unless elevated due to Gilbert's syndrome)
   * ALT/AST ≤ 2.5 x ULN (≤ 5 x ULN for participants with known hepatic metastases)
10. Participants must have adequate renal function based on the following:

    * Serum creatinine ≤ 1.5 x ULN; or
    * Serum creatinine clearance ≥ 60 mL/min, as determined by Cockcroft-Gault equation
11. For women of childbearing potential (WCBP): negative urine pregnancy test (UPT) within 1 week before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 12 consecutive months for women > 55 years of age). WCBP should be placed on effective birth control directly after testing negative for pregnancy; if not, then WCBP should have a UPT on Day 1 of every cycle, prior to study intervention administration. Any positive or indeterminant UPT result must be confirmed by serum.

    a. Female participants of childbearing potential must use a highly effective mode of contraception or abstain from heterosexual activity for the duration of the study and for 120 days following the last dose of study intervention. A female is NOT of childbearing potential if she has undergone bilateral salpingoophorectomy or is menopausal, defined as an absence of menses for 12 consecutive months. Male participants must agree to use highly effective contraception.
12. Ability to adhere to the study visit schedule and all protocol requirements
13. Must be able to swallow capsules

Participants will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

Participants are to be excluded from the study if they meet any of the following criteria:

1. Major surgery within 4 weeks prior to Screening
2. Participants with active CNS metastases; however, participants who have undergone radiation and/or surgery for the treatment of CNS metastases, who are neurologically stable and who are no longer taking pharmacologic doses of corticosteroids are eligible; participants with leptomeningeal metastases are not eligible.
3. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
4. Prior anti-cancer therapy within 4 weeks prior to the start of study intervention. A 2 week washout is acceptable for short-acting drugs (eg, tyrosine kinase inhibitors). Any treatment-related toxicities must be resolved to Grade 0 - 1.
5. Human immunodeficiency virus (HIV)-infected participants
6. Participants who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment.

   Note: Participants should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.

   Hepatitis B screening tests are not required unless:
   * Known history of HBV infection
   * As mandated by local health authority
7. Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at Screening. Note: Participants must have completed curative antiviral therapy at least 4 weeks prior to enrollment.

   Hepatitis C screening tests are not required unless:
   * Known history of HCV infection
   * As mandated by local health authority
8. Participants who require immunosuppressive therapy including, but not limited to, treatment with corticosteroids in pharmacologic doses (equivalent to ≥ 10 mg prednisone daily), cyclosporine, mycophenolate, azathioprine, methotrexate, adalimumab, infliximab, vedolizumab, tofacitinib, dupilumab, rituximab, etc. or systemic steroids (except for steroid use as cortisol replacement therapy in documented adrenal insufficiency)
9. Participants requiring administration of drugs known to be strong inhibitors or inducers of CYP3A4, 2C9 or 2C19
10. Participants requiring drugs that modify gastric pH, such as proton-pump inhibitors (PPIs) or H2 blockers. Antacids, such as calcium carbonate or aluminum hydroxide-based products, will be allowed during the study, but are recommended to be taken either 4 hours before or 2 hours after dosing of TT 10 (PORT 6) or PORT-7.
11. Ongoing systemic bacterial, fungal or viral infections at Screening

    a. NOTE: Participants on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met
12. Administration of a live vaccine within 6 weeks of first dose of study intervention. Messenger ribonucleic acid (mRNA) vaccines for the prevention of Coronavirus Disease 2019 (COVID-19) infection are permitted.
13. Baseline QT interval corrected with Fridericia's method (QTcF) > 470 ms (average of triplicate readings)

    a. NOTE: Criterion does not apply to participants with a right or left bundle branch block.
14. Prior surgery or gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy)
15. Female participants who are pregnant or breastfeeding
16. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix or prostate intraepithelial neoplasia
17. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
18. History of peptic ulcer and/or gastrointestinal bleed within the past 6 months prior to Screening
19. History of stroke, unstable angina, myocardial infarction or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening
20. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the participant associated with his or her participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Dose Limiting Toxicities (DLTs) of TT-10, TT-4 and TT-10 + TT-4 during the dose escalation phase | 28 Days
  All toxicities will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Define the maximum tolerated dose (MTD) or phase 2 recommended dose of TT-10, TT-4 and TT-10 + TT-4 during the dose escalation phase | Through study completion, an average of 1 year
  To confirm the maximum tolerated dose (MTD) of TT-10, TT-4 and TT-10 + TT-4, defined as the highest dose level at which <2 out of 6 participants experience a dose-limiting toxicity
Expansion cohort primary objective - safety | Through study completion, an average of 1 year
  Incidence and severity of treatment-related adverse events (TRAEs) in participants treated at the recommended phase 2 dose in the expansion phase

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  ORR is to be reported as the proportion of patients who have a Complete Response or Partial Response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Duration of Response (DoR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  Defined as the time from first documented objective response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 to the date of first documented radiographic progression of disease (PD) or death.
Progression Free Survival (PFS) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  Time from first dose to the date of the first confirmed documented progression per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Peak serum concentration (Cmax) of TT-10 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter
Area under the serum concentration versus time curve (AUC) of TT-10 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter
Half-life of TT-10 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Norton Cancer Institute, Louisville, Kentucky
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang J, Yan W, Duan W, Wuthrich K, Cheng J. Tumor Immunotherapy Using A2A Adenosine Receptor Antagonists. Pharmaceuticals (Basel). 2020 Sep 8;13(9):237. doi: 10.3390/ph13090237. PMID 32911819
- [Background] Allard B, Allard D, Buisseret L, Stagg J. The adenosine pathway in immuno-oncology. Nat Rev Clin Oncol. 2020 Oct;17(10):611-629. doi: 10.1038/s41571-020-0382-2. Epub 2020 Jun 8. PMID 32514148
- [Background] Beavis PA, Henderson MA, Giuffrida L, Mills JK, Sek K, Cross RS, Davenport AJ, John LB, Mardiana S, Slaney CY, Johnstone RW, Trapani JA, Stagg J, Loi S, Kats L, Gyorki D, Kershaw MH, Darcy PK. Targeting the adenosine 2A receptor enhances chimeric antigen receptor T cell efficacy. J Clin Invest. 2017 Mar 1;127(3):929-941. doi: 10.1172/JCI89455. Epub 2017 Feb 6. PMID 28165340
- [Background] Willingham SB, Hotson AN, Miller RA. Targeting the A2AR in cancer; early lessons from the clinic. Curr Opin Pharmacol. 2020 Aug;53:126-133. doi: 10.1016/j.coph.2020.08.003. Epub 2020 Sep 29. PMID 33002857
- [Background] Vijayan D, Young A, Teng MWL, Smyth MJ. Targeting immunosuppressive adenosine in cancer. Nat Rev Cancer. 2017 Dec;17(12):709-724. doi: 10.1038/nrc.2017.86. Epub 2017 Oct 23. PMID 29059149
- [Background] Steingold JM, Hatfield SM. Targeting Hypoxia-A2A Adenosinergic Immunosuppression of Antitumor T Cells During Cancer Immunotherapy. Front Immunol. 2020 Sep 29;11:570041. doi: 10.3389/fimmu.2020.570041. eCollection 2020. PMID 33117358
- [Background] Sek K, Molck C, Stewart GD, Kats L, Darcy PK, Beavis PA. Targeting Adenosine Receptor Signaling in Cancer Immunotherapy. Int J Mol Sci. 2018 Dec 2;19(12):3837. doi: 10.3390/ijms19123837. PMID 30513816
- [Background] Vigano S, Alatzoglou D, Irving M, Menetrier-Caux C, Caux C, Romero P, Coukos G. Targeting Adenosine in Cancer Immunotherapy to Enhance T-Cell Function. Front Immunol. 2019 Jun 6;10:925. doi: 10.3389/fimmu.2019.00925. eCollection 2019. PMID 31244820
- [Background] Schwarzacher SW, Krammer EB. Complex anomalies of the human aortic arch system: unique case with both vertebral arteries as additional branches of the aortic arch. Anat Rec. 1989 Nov;225(3):246-50. doi: 10.1002/ar.1092250310. PMID 2817442
- [Background] Helms RS, Powell JD. Rethinking the adenosine-A2AR checkpoint: implications for enhancing anti-tumor immunotherapy. Curr Opin Pharmacol. 2020 Aug;53:77-83. doi: 10.1016/j.coph.2020.07.003. Epub 2020 Aug 9. PMID 32781414
- [Background] Kamai T, Kijima T, Tsuzuki T, Nukui A, Abe H, Arai K, Yoshida KI. Increased expression of adenosine 2A receptors in metastatic renal cell carcinoma is associated with poorer response to anti-vascular endothelial growth factor agents and anti-PD-1/Anti-CTLA4 antibodies and shorter survival. Cancer Immunol Immunother. 2021 Jul;70(7):2009-2021. doi: 10.1007/s00262-020-02843-x. Epub 2021 Jan 8. PMID 33416945
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869